CLINICAL TRIAL: NCT00635427
Title: An Open-Label Extension Study of Gene-Activated® Human Glucocerebrosidase (GA-GCB) Enzyme Replacement Therapy in Patients With Type 1 Gaucher Disease
Brief Title: An Open-Label Extension Study of GA-GCB ERT in Patients With Type 1 Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-GCB-044; 2008-001965-27 (EudraCT Number)
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2014-01-28 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Gaucher Disease, Type 1
Keywords: VPRIV; Enzyme Replacement Therapy; Gaucher disease; glucocerebrosidase; beta-glucocerebrosidase; Acid beta-glucocerebrosidase; glucosylceramidase; D-glucosyl-N-acylsphingosine glucohydrolase; gene activation; human
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- VPRIV 60 U/kg(VPRIV Parent Study 45 or 60 U/kg- TKT032,GCB039) (Experimental): This arm is the Overall velaglucerase alfa (VPRIV) 60 U/kg and includes patients from the following groups:
  VPRIV 45 U/kg or 60 U/kg, IV, EOW for 51 weeks in parent study TKT032 (NCT00430625) and switched to 60 U/kg in HGT-GCB-044 to maintain blindness or 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631)
  Interventions: Biological: VPRIV®
- VPRIV 60 U/kg (Parent study-imiglucerase(60 U/kg) HGT-GCB-039) (Experimental): imiglucerase 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631)and switched 60 U/kg VPRIV in HGT-GCB-044
  Interventions: Biological: VPRIV®
- VPRIV 15-60 U/kg (Parent study VPRIV (15-60 U/kg) TKT034) (Experimental): VPRIV 15- 60 U/kg, IV, EOW for 51 weeks in parent study TKT034 (NCT00478647) and continued in HGT-GCB-044 at the same dose as prescribed in TKT034
  Interventions: Biological: VPRIV®

INTERVENTIONS:
Biological: VPRIV® — Intravenous infusion, every other week (EOW)
  Other Names: velaglucerase alfa; Gene-Activated® Human Glucocerebrosidase(GA-GCB)

SUMMARY:
The purpose of this study is to evaluate the long-term safety of every other week dosing of Gene-Activated® human glucocerebrosidase (GA-GCB, velaglucerase alfa) intravenously in patients with type 1 Gaucher disease.

DETAILED DESCRIPTION:
Type 1 Gaucher disease, the most common form,accounts for more than 90% of all cases and does not involve the CNS. Typical manifestations of type 1 Gaucher disease include hepatomegaly, splenomegaly, thrombocytopenia, bleeding tendencies, anemia, hypermetabolism, skeletal pathology, growth retardation, pulmonary disease, and decreased quality of life. Gene-Activated® human glucocerebrosidase (GA-GCB,velaglucerase alfa) is produced in a continuous human cell line using proprietary gene-activation technology and has an identical amino acid sequence to the naturally occurring human enzyme. GA-GCB contains terminal mannose residues that target the enzyme to the macrophages-the primary target cells in Gaucher disease. This study was designed to determine the long-term safety of GA-GCB in men, women, and children with Type 1 Gaucher disease.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has completed study TKT032 or TKT034, or study HGT-GCB-039.
2. Female patients of child-bearing potential must agree to use a medically acceptable method of contraception at all times during the study and must have negative results to a pregnancy test performed at the time of enrollment and as required throughout their participation in the study.
3. Male patients must agree to use a medically acceptable method of contraception at all times during the study and report a partner's pregnancy to the investigator.
4. The patient, the patient's parent(s) or legal guardian(s) has provided written informed consent that has been approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC).
5. The patient must be sufficiently cooperative to participate in this clinical study as judged by the Investigator

Exclusion Criteria:

1. The patient has received treatment with any non-Gaucher disease-related investigational drug or device within the 30 days prior to study entry; such use during the study is not permitted.
2. The patient is pregnant or lactating.
3. The patient, patient's parent(s), or patient's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study.
4. The patient has a significant comorbidity(ies) that might affect study data or confound the study results (e.g., malignancies, primary biliary cirrhosis, autoimmune liver disease, etc.).
5. The patient is unable to comply with the protocol, e.g., has a clinically relevant medical condition making implementation of the protocol difficult, has an uncooperative attitude, is unable to return for safety evaluations, or is otherwise unlikely to complete the study, as determined by the Investigator

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-03-13 (Actual); Primary Completion 2012-12-28 (Actual); Study Completion 2012-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (21):
- United States (10):
  - Los Angeles Medical Center, Los Angeles, California
  - Children's Hospital Oakland, Oakland, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - NYU Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah Medical Center, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Your Health S.A., Buenos Aires, Argentina
- India (2):
  - All India Institute of Medical Sciences, New Delhi
  - KEM Hospital, Pune
- Shaare Zedek Medical Center, Jerusalem, Israel
- Sociedad Espanola de Socorros Mutuos, Asunción, Paraguay
- Instytut "Pomnik-Centrum Zdrowia Dziecka", Warsaw, Poland
- State Institution "Hematology Research Centre RAMS", Moscow, Russia
- Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do, South Korea
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- Hospital de La Rabta, Tunis, Jebbari, Tunisia
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] Zimran A, Elstein D, Gonzalez DE, Lukina EA, Qin Y, Dinh Q, Turkia HB. Treatment-naive Gaucher disease patients achieve therapeutic goals and normalization with velaglucerase alfa by 4years in phase 3 trials. Blood Cells Mol Dis. 2018 Feb;68:153-159. doi: 10.1016/j.bcmd.2016.10.007. Epub 2016 Oct 21. PMID 27839979
- [Derived] Smith L, Rhead W, Charrow J, Shankar SP, Bavdekar A, Longo N, Mardach R, Harmatz P, Hangartner T, Lee HM, Crombez E, Pastores GM. Long-term velaglucerase alfa treatment in children with Gaucher disease type 1 naive to enzyme replacement therapy or previously treated with imiglucerase. Mol Genet Metab. 2016 Feb;117(2):164-71. doi: 10.1016/j.ymgme.2015.05.012. Epub 2015 Jun 1. PMID 26043810
- [Derived] Hughes DA, Gonzalez DE, Lukina EA, Mehta A, Kabra M, Elstein D, Kisinovsky I, Giraldo P, Bavdekar A, Hangartner TN, Wang N, Crombez E, Zimran A. Velaglucerase alfa (VPRIV) enzyme replacement therapy in patients with Gaucher disease: Long-term data from phase III clinical trials. Am J Hematol. 2015 Jul;90(7):584-91. doi: 10.1002/ajh.24012. PMID 25801797

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled in the study on 13 March 2008 and the last participant completed study procedures on 28 December 2012.
Pre-assignment Details: 2 participants who did not have type 1 Gaucher disease were withdrawn from the intent-to-treat (ITT) set as per the statistical analysis plan and removed from the long-term efficacy analyses in this study, needed to support the interpretation of the long-term efficacy results. Hence, 93 of 95 participants were included in the HGT-GCB-044 ITT set.
Groups:
- VPRIV 60 U/kg (Parent Study VPRIV (45 U/kg) -TKT032): VPRIV 45 U/kg, IV, every other week (EOW) for 51 weeks in parent study TKT032 (NCT00430625) and switched to 60 U/kg in HGT-GCB-044
- VPRIV 60 U/kg (Parent Study- VPRIV (60 U/kg)-TKT032): VPRIV 60 U/kg, IV, EOW for 51 weeks in parent study TKT032 (NCT00430625)
- VPRIV 60 U/kg (Parent Study- VPRIV (60U/kg) HGT-GCB-039): VPRIV 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631)
- VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg)HGT-GCB-039): imiglucerase 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631)and switched 60 U/kg VPRIV in HGT-GCB-044
- VPRIV 15-60 U/kg (Parent Study VPRIV(15-60 U/kg)TKT034): VPRIV 15- 60 U/kg, IV, EOW for 51 weeks in parent study TKT034 (NCT00478647) and continued in HGT-GCB-044 at the same dose as prescribed in TKT034
Period: Overall Study
Arm/Group | VPRIV 60 U/kg (Parent Study VPRIV (45 U/kg) -TKT032) | VPRIV 60 U/kg (Parent Study- VPRIV (60 U/kg)-TKT032) | VPRIV 60 U/kg (Parent Study- VPRIV (60U/kg) HGT-GCB-039) | VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg)HGT-GCB-039) | VPRIV 15-60 U/kg (Parent Study VPRIV(15-60 U/kg)TKT034)
Started | 13 (12 participants were considered ITT population as 1 participant did not have type 1 Gaucher disease) | 12 (11 participants were considered ITT population as 1 participant did not have type 1 Gaucher disease) | 16 | 16 | 38
Completed | 1 | 6 | 5 | 7 | 30
Not Completed | 12 | 6 | 11 | 9 | 8
Not completed — Refusal Of Required DiagnosticEvaluation | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Termination Of Study By Sponsor | 12 | 6 | 10 | 6 | 6
Not completed — Withdrawal Of Consent | 0 | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Two participants who did not have type 1 Gaucher disease were withdrawn from the ITT study as per SAP definition and removed from the long-term efficacy analyses in this study, needed to support the interpretation of the long-term efficacy results. Therefore, 93 of 95 (97.9%) participants were included in the HGT-GCB-044 ITT population.
Groups:
- VPRIV 60 U/kg (Parent Study VPRIV (45 U/kg)-TKT032): VPRIV 45 U/kg, IV, EOW for 51 weeks in parent study TKT032 (NCT00430625) and switched to 60 U/kg in HGT-GCB-044.
- VPRIV 60 U/kg (Parent Study VPRIV (60 U/kg)-TKT032): VPRIV 60 U/kg, IV, EOW for 51 weeks in parent study TKT032 (NCT00430625).
- VPRIV 60 U/kg (Parent Study VPRIV (60U/kg) HGT-GCB-039): VPRIV 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631).
- VPRIV 60 U/kg (Parent Study-imiglucerase (60 U/kg) HGT-GCB-039: Imiglucerase 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631) and switched 60 U/kg VPRIV in HGT-GCB-044
- VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034): VPRIV 15- 60 U/kg, IV, EOW for 51 weeks in parent study TKT034 (NCT00478647). Participants continued to receive VPRIV at a dose of 15-60 U/kg throughout participation in HGT-GCB-044
- Total: Total of all reporting groups
Arm/Group | VPRIV 60 U/kg (Parent Study VPRIV (45 U/kg)-TKT032) | VPRIV 60 U/kg (Parent Study VPRIV (60 U/kg)-TKT032) | VPRIV 60 U/kg (Parent Study VPRIV (60U/kg) HGT-GCB-039) | VPRIV 60 U/kg (Parent Study-imiglucerase (60 U/kg) HGT-GCB-039 | VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034) | Total
Number analyzed (Participants) | 12 | 11 | 16 | 16 | 38 | 93
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time the informed consent was obtained in the core study.
  Years | 32.5 (16.75) | 22 (11.08) | 32.9 (16.14) | 25 (17.33) | 34.3 (17.94) | 31.4 (17.15)
Age, Customized [Count of Participants; unit: Participants] — Age at the time the informed consent was obtained in the core study.
  Participants
    At least 18 years | 2 | 3 | 3 | 5 | 9 | 22
    Between 18 and 65 years | 10 | 8 | 13 | 11 | 26 | 68
    Greater than or equal to 65 years | 0 | 0 | 0 | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 8 | 7 | 18 | 46
  Male | 5 | 5 | 8 | 9 | 20 | 47
Splenectomy status [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 9 | 10 | 3 | 22
  No | 12 | 11 | 7 | 6 | 35 | 71
Baseline hemoglobin concentration per treatment group [Mean (Full Range); unit: gram per deciliter] — Baseline was defined as data collected prior to the first dose in the core study (TKT032, TKT034, and HGT-GCB-039).
  gram per deciliter | 10.68 [8.5 to 12.9] | 10.68 [7.1 to 12.3] | 11.56 [9.7 to 14.4] | 10.58 [8.1 to 13.1] | 13.82 [10.7 to 16.5] | 12.09 [7.1 to 16.5]
Baseline platelet counts per treatment group [Mean (Full Range); unit: x10^9/L] — Baseline was defined as data collected prior to the first dose in the core study (TKT032, TKT034, and HGT-GCB-039).
  x10^9/L | 69.3 [13 to 146] | 79.4 [47 to 139] | 160.1 [44 to 310] | 186.3 [63 to 430] | 165.4 [29 to 399] | 144.81 [13 to 430]
Baseline liver volume per treatment group [Mean (Full Range); unit: Percent (%) body weight] — Baseline was defined as data collected prior to the first dose in the core study (TKT032, TKT034, and HGT-GCB-039). Normal liver volume was defined as 2.5 percent of body weight.
  Percent (%) body weight | 1.64 [1.1 to 2.9] | 1.63 [1 to 3.2] | 1.59 [0.8 to 2.2] | 1.68 [0.7 to 2.8] | 0.82 [0.6 to 1.3] | 1.302 [0.6 to 3.2]
Baseline Spleen volume per treatment group [Mean (Full Range); unit: Multiple of Normal] — Baseline was defined as data collected prior to the first dose in the core study (TKT032, TKT034, and HT-GCB-039). Normal spleen volume is defined as 0.2 percentage of body weight.
  Multiple of Normal | 23.08 [4.8 to 65.1] | 18.48 [5.7 to 36.9] | 12.69 [7.2 to 31.6] | 23.52 [3.1 to 44.4] | 4.1 [1.2 to 15.8] | 13.07 [1.2 to 65.1]

OUTCOME MEASURES:

1. Primary Outcome: Overall Summary of Treatment Emergent Adverse Events
Description: Safety was evaluated by an analysis of adverse events (AEs), concomitant medication use, clinical laboratory tests, vital signs during the infusion of study drug, physical examination, and the development of anti-velaglucerase alfa. No formal comparisons or statistical tests were applied for the safety analyses, including for differences between the groups.
Time Frame: Baseline to termination of study
Population: All participants who received at least 1 infusion (full or partial) of study drug were evaluated for safety (ie, were included in the safety population). There were 95 participants in the safety population.
Measure: Number; unit: Participants
Groups:
- VPRIV 60 U/kg(Parent Study VPRIV(45 or 60 U/kg) TKT032,GCB039): This is the overall velaglucerase alfa group consisting of the following population: VPRIV 45 U/kg or 60 U/kg, IV, EOW for 51 weeks in parent study TKT032 (NCT00430625) and switched to 60 U/kg in HGT-GCB-044 to maintain blindness or 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631)
- VPRIV 60 U/kg (Parent Study-imiglucerase (60 U/kg)HGT-GCB-039): imiglucerase 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631)and switched to 60 U/kg VPRIV in HGT-GCB-044
Arm/Group | VPRIV 60 U/kg(Parent Study VPRIV(45 or 60 U/kg) TKT032,GCB039) | VPRIV 60 U/kg (Parent Study-imiglucerase (60 U/kg)HGT-GCB-039) | VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034)
Number analyzed (Participants) | 41 | 16 | 38
Participants
  Experienced no AEs | 3 | 1 | 3
  Experienced at least 1 AE | 38 | 15 | 35
  Experienced at least 1 drug-related AE | 9 | 7 | 8
  Experienced at least 1 infusion-related AE | 5 | 1 | 5
  Experienced at least 1 severe AE | 4 | 3 | 4
  Experienced at least 1 drug-related severe AE | 0 | 0 | 0
  Experienced at least 1 Life-threatening AE | 0 | 0 | 0
  Experienced at least 1 drug-related Life-threateni | 0 | 0 | 0
  Experienced at least 1 serious AE | 6 | 4 | 6
  Experienced at least 1 drug-related serious AE | 0 | 0 | 0
  Discontinued due to an AE | 0 | 0 | 0
  Deaths | 0 | 1 | 0

2. Secondary Outcome: Change From Baseline to 24 Months in Hemoglobin Concentration for Each Treatment Group
Time Frame: Baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: (g/dL)
Groups:
- VPRIV 60 U/kg(VPRIV Parent Study 45 or 60 U/kg- TKT032,GCB039): This arm is the Overall velaglucerase alfa (VPRIV) 60 U/kg and includes participants from the following groups: VPRIV 45 U/kg or 60 U/kg, IV, EOW for 51 weeks in parent study TKT032 (NCT00430625) and switched to 60 U/kg in HGT-GCB-044 to maintain blindness or 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631)
- VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg) HGT-GCB-039): imiglucerase 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631)and switched to 60 U/kg VPRIV in HGT-GCB-044
Arm/Group | VPRIV 60 U/kg(VPRIV Parent Study 45 or 60 U/kg- TKT032,GCB039) | VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg) HGT-GCB-039) | VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034)
Number analyzed (Participants) | 39 | 16 | 38
(g/dL) | 2.75 [2.28 to 3.22] | 2.00 [1.25 to 2.75] | -0.05 [-0.34 to 0.25]

3. Secondary Outcome: Change From Baseline to 24 Months in Platelet Counts for Each Treatment Group
Time Frame: Baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: (10^9/L)
Arm/Group | VPRIV 60 U/kg(VPRIV Parent Study 45 or 60 U/kg- TKT032,GCB039) | VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg) HGT-GCB-039) | VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034)
Number analyzed (Participants) | 39 | 16 | 38
(10^9/L) | 87.85 [72.69 to 103.00] | 160.94 [117.22 to 204.66] | 9.03 [-2.60 to 20.66]

4. Secondary Outcome: Change From Baseline to 24 Months in Normalized Liver Volume for Each Treatment Group
Time Frame: Baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: % Body weight
Arm/Group | VPRIV 60 U/kg(VPRIV Parent Study 45 or 60 U/kg- TKT032,GCB039) | VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg) HGT-GCB-039) | VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034)
Number analyzed (Participants) | 39 | 16 | 38
% Body weight | -1.206 [-1.501 to -0.912] | -1.688 [-2.164 to -1.211] | -0.026 [-0.100 to 0.047]

5. Secondary Outcome: Percentage Change From Baseline to 24 Months in Normalized Spleen Volume for Each Treatment Group
Time Frame: Baseline to 24 months
Measure: Mean (95% Confidence Interval); unit: Precent (%) change
Arm/Group | VPRIV 60 U/kg(VPRIV Parent Study 45 or 60 U/kg- TKT032,GCB039) | VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg) HGT-GCB-039) | VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034)
Number analyzed (Participants) | 39 | 16 | 38
Precent (%) change | -64.49 [-69.26 to -59.73] | -63.82 [-89.65 to -37.98] | -8.04 [-14.00 to -2.08]

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were defined as AEs which occurred on or after the time of the first infusion in HGT-GCB-044, until 30 days after the participant's last study infusion.
Description: AEs may have been discovered through observation or examination, and questioning of the participant, complaint by the participant, or by an abnormal clinical laboratory value. Severity of AEs was to be assessed by the investigator and recorded on the electronic case report form (eCRF)regardless of the severity or relationship to study drug.
Groups:
- VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg) HGT-GCB-039): imiglucerase 60 U/kg, IV, EOW for 39 weeks in parent study HGT-GCB-039 (NCT00553631) and switched 60 U/kg VPRIV in HGT-GCB-044
Arm/Group | VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034) | VPRIV 60 U/kg(VPRIV Parent Study 45 or 60 U/kg- TKT032,GCB039) | VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg) HGT-GCB-039)
Serious Adverse Events (participants affected / at risk) | 6/38 | 6/41 | 4/16
Other Adverse Events (participants affected / at risk) | 35/38 | 35/41 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034) (N=38) | VPRIV 60 U/kg(VPRIV Parent Study 45 or 60 U/kg- TKT032,GCB039) (N=41) | VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg) HGT-GCB-039) (N=16)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (3)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VPRIV 15-60 U/kg (Parent Study VPRIV (15-60 U/kg) TKT034) (N=38) | VPRIV 60 U/kg(VPRIV Parent Study 45 or 60 U/kg- TKT032,GCB039) (N=41) | VPRIV 60 U/kg (Parent Study-imiglucerase(60 U/kg) HGT-GCB-039) (N=16)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 4 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (4) | 3 (3) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (3) | 6 (7) | 2 (2)
Fatigue (General disorders) | 7 (8) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 6 (10) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 5 (13) | 1 (1)
Bronchitis acute (Infections and infestations) | 0 (0) | 5 (5) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 7 (10) | 1 (1)
Influenza (Infections and infestations) | 4 (6) | 6 (10) | 4 (12)
Nasopharyngitis (Infections and infestations) | 16 (31) | 11 (20) | 3 (4)
Pharyngitis (Infections and infestations) | 5 (11) | 2 (2) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 4 (13) | 1 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 4 (7) | 6 (14)
Urinary tract infection (Infections and infestations) | 3 (5) | 3 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 14 (33) | 2 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 5 (6) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (12) | 7 (20) | 2 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 5 (6) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (4) | 1 (2)
Headache (Nervous system disorders) | 6 (10) | 7 (16) | 4 (6)
Paraesthesia (Nervous system disorders) | 2 (2) | 2 (2) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0) | 3 (4)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 4 (6) | 5 (6) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 2 (3) | 0 (0) | 0 (0)
Dental caries (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hepatitis a (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 2 (3)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 3 (5) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Hyperprolactinaemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 1 (3)
Drop attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Haematoma (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Lentigo (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Galactorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (6) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Aspartate aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood creatine phosphokinase Increased (Investigations) | 2 (2) | 1 (3) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Mean cell volume increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 2 (2) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (7)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 3 (6) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Shire's agreements with investigators vary. All agreements provide Shire the right to embargo communications regarding trial results prior to public release for a period ≤180 days from the time submitted to Shire for review. Shire does not prohibit publication, but can require the removal of confidential information(excluding trial results) and can request postponement of a single-center publication until after disclosure of the trial's multi-center publication